CLINICAL TRIAL: NCT00119405
Title: Role of Mitochondria in the Development of HIV Atrophy
Brief Title: Observational Study of Fat Loss in HIV Infected Adults Taking Nucleoside Reverse Transcriptase Inhibitors (NRTIs)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01AI060484-01A2A; 1R01-AI060484-01A2A; 1R01AI060484-01A2 (NIH)
Record Dates: First submitted 2005-07-11; First posted 2005-07-13 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2007-12

CONDITIONS: HIV Infections; Lipodystrophy; Metabolic Diseases; Nutrition Disorders
Keywords: Lipoatrophy; Mitochondria; Treatment Naive
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Metabolic Diseases; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fat and Blood for mitochindrial DNA and different nuclear genes that regulate fat and lipid metabolism
Oversight: Data Monitoring Committee: No

SUMMARY:
Nucleoside reverse transcriptase inhibitors (NRTIs) are a class of anti-HIV (Human Immunodeficiency Virus) drug that can be an important part of an HIV treatment regimen. Because anti-HIV therapy may have negative side effects, there is a great need to carefully study HIV infected patients on such regimens. One negative side effect observed in many HIV infected patients is lipoatrophy, a condition that results in fat loss in the body. It is unclear if NRTIs also have a role in the development of mitochondrial toxicity, a condition that affects the body's ability to produce energy. The purpose of this study is to observe the effects of an NRTI-based, protease inhibitor (PI)-sparing drug regimen on fat loss in HIV infected, treatment-naive adults.

Study hypothesis: The initiation of NRTI-containing, PI-sparing therapy will inhibit mitochondrial DNA (mtDNA) synthesis and lead to a decrease in mtDNA content in adipose tissue, skeletal muscle and peripheral blood mononuclear cells (PBMCs), will cause deterioration in mitochondrial function, will increase fat apoptosis and oxidative damage biomarkers, and will lead to progressive decrease in body fat content.

DETAILED DESCRIPTION:
NRTIs are a mainstay of HIV treatment regimens, often part of initial treatment regimens for newly diagnosed patients. Recent data suggest that NRTIs are responsible for lipoatrophy, a condition marked by progressive fat loss. Another negative side effect to antiretroviral (ARV) regimens is mitochondrial toxicity, which can damage the heart, nerves, muscles, kidneys, pancreas and liver, as well as affecting the body's ability to produce energy for important life processes. It has been hypothesized that lipoatrophy may be related to mitochondrial toxicity, but a causal relationship between the two has yet to be established. This study will examine HIV infected treatment-naive patients who are initiating their first ARV regimens. The regimens will contain 2 NRTI, one of which being zidovudine and a non-nucleoside reverse transcriptase inhibitor (NNRTI). The regimens will not contain any PIs.

Patients will participate in this study for 96 weeks. There will be 4 study visits at Weeks 12, 24, 48, and 96. Dual-energy x-ray absorptiometry (DEXA) scans and fat biopsies will occur at all visits. Additionally, blood collection for metabolic testing will occur at Week 12. ARVs will not be provided by this study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Treatment-naive
* Plan to initiate first ARV regimen with 2 NRTIs and an NNRTI
* Plan to include zidovudine as part of first ARV regimen

Exclusion Criteria:

* Current use of steroids or growth hormone
* Coagulopathies or other bleeding disorders
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive adults starting their first antiretroviral regimen with either azidothymidine (AZT)-containing combination
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2005-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace A. McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 6/2005 to 11/2008. Participants were recruited from 3 HIV clinics in Cleveland, with the majority from the clinic at University Hospitals Case Medical Center.
Pre-assignment Details: Participants had to be HIV+ and naive to ARVs.
Groups:
- ARV Naive: ARV naive
Period: Overall Study
Arm/Group | ARV Naive
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ARV Naive
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.88 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Mitochondrial Function (mtDNA Levels)
Description: Mitochondrial gene expression: mtDNA levels are used to quantify this outcome measure.
Time Frame: 96 weeks
Measure: Mean (95% Confidence Interval); unit: copies per cell
Groups:
- ARV Naive: ARV naive (have never been on antiretrovirals before)
Arm/Group | ARV Naive
Number analyzed (Participants) | 18
copies per cell | 1372 [532 to 2721]

ADVERSE EVENTS:
Arm/Group | ARV Naive
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARV Naive (N=18)
Pancreatitis (Grade 3) (Endocrine disorders) | 1 (1)
Right Lower Lobe (RLL) Pneumonia (Grade 3) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Grade 2) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARV Naive (N=18)
Incisional Seroma (Skin and subcutaneous tissue disorders) | 1 (1)
Incisional Hematoma (Grade 1) (Skin and subcutaneous tissue disorders) | 2 (2)
Infected Incisional Hematoma (Grade 2) (Skin and subcutaneous tissue disorders) | 1 (1)
Low glucose 34 (Grade 3) (Metabolism and nutrition disorders) | 1 (1) — Lab delay - repeated result was 105
Low glucose 48 (Grade 2) (Metabolism and nutrition disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Grade 2) (Cardiac disorders) | 1 (1)
Bone Mineral Density (BMD)/T scores -2.3 and -3.2 (Musculoskeletal and connective tissue disorders) | 1 (1) — Known osteoporosis pre-study
Elevated Aspartate aminotransferase (AST) (Grades 2 and 3) (Hepatobiliary disorders) | 3 (3)
Elevated creatine kinase (CK) levels (Grades 3 and 4) (Musculoskeletal and connective tissue disorders) | 3 (3)
Elevated alanine aminotransferase (ALT) 207 (Grade 2) (Hepatobiliary disorders) | 1 (1)
Elevated Cholesterol 257 (Grade 2) (Metabolism and nutrition disorders) | 1 (1)
Elevated low-density lipoprotein (LDL) 175 (Grade 2) (Metabolism and nutrition disorders) | 1 (1)
Low absolute neutrophil count (ANC) (Grades 2 and 3) (Blood and lymphatic system disorders) | 2 (3)
Low white blood cell (WBC) count (Grade 2) (Blood and lymphatic system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes